CLINICAL TRIAL: NCT02390206
Title: An Observational, Prospective, Multicentre, National Trial on the Benefit of Botulinum Toxin Type A (BoNT-A) Injections in Untreated Chronic Post-stroke Spastic Brazilian Patients
Brief Title: Study on the Use of Botulinum Toxin Type A in the Treatment of Chronic Post-stroke Spastic Patients
Acronym: B-CAUSE
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-38-52120-202
Record Dates: First submitted 2015-03-04; First posted 2015-03-17 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Spasticity
Keywords: Stroke; Spasticity; Botulinum Toxin type A; Dysport
MeSH Terms: conditions — Muscle Spasticity; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Botulinum toxin type A (BoNT-A) injection Naïve: Subjects naïve to BoNT-A treatment. Investigators follow their individual injection protocol for treatment with BoNT-A (modalities of administration in accordance with local Summary of Product Characteristics and locally agreed therapeutic guidelines).

SUMMARY:
The purpose of this study is to document the effectiveness of treating chronic post-stroke spastic patients with Botulinum Toxin type A.

DETAILED DESCRIPTION:
As this is a non-interventional study, the decision to prescribe the product must be taken prior to, and independently from the decision to enrol the patient. This decision should be made in accordance with routine clinical practice at the hospital concerned. The clinical justification for prescribing any treatment should be recorded at the outset by the prescribing clinician.

This study will not interfere with the routine practice of the investigator or with the patient's treatment plan. Assessments will be done only if performed regularly in routine practice.

This study will be conducted in Brazil, wherein Marketing Authorization has been granted for the use of BoNT-A in the treatment of spasticity of the upper and lower limb in adult post-stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Time between last documented stroke (either haemorrhagic or ischemic) and study inclusion date equal or longer than 1 year
* Documented upper limb spasticity, with or without lower limb spasticity
* Naive to BoNT-A injections for spasticity treatment
* Provide written informed consent (signed by the patient or his legal representative) prior to any study-related procedure

Exclusion Criteria:

* Previous surgical procedure for spasticity treatment, including neurotomy, rhizotomy and intrathecal pump implants
* Previous phenol injection and/or indication to receive phenol during the study duration
* Contraindications to any BoNT-A preparations
* Patient and/or caregiver unable to comply with the study requirements
* The patient has already been included in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Untreated chronic post-stroke spastic patients
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2015-06; Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Change in Goal Achievement Score (GAS). | 3 and 6 months

SECONDARY OUTCOMES:
Change from baseline in pain according to Verbal Numerical Scale (VNS). | Baseline and 3 months
Change from baseline in Modified Ashworth Scale (MAS) score | Baseline and 3 months
Change from baseline in functional independence according to Barthel index score | Baseline and 3 months
Change from baseline in Quality of Life according to Euro-5D-5L health questionnaire | Baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (11):
- Brazil (11):
  - Hospital Bettina Ferro de Souza Campus IV da Universidade Federal do Pará, Belém
  - Centro Catarinense de Reabilitação, Florianópolis
  - Centro de Reabilitação e Readaptação Dr. Henrique Santillo, Goiânia
  - Clinica Neurológica e Neurocirúrgica de Joinville, Joinville
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto
  - Hospital Universitário Clementino Fraga Filho (HUCFF), Rio de Janeiro
  - Instituto de Reabilitação Lucy Montoro - FAMERP, São José do Rio Preto
  - Irmandade da Santa Casa de Misericórida de São Paulo, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo
  - Hospital São Paulo - UNIFESP, São Paulo
  - HCSP - Complexo Hospital das Clinicas Instituto de Medicina Fisica e Reabilitação, São Paulo